CLINICAL TRIAL: NCT05084495
Title: Can Global Peak Longitudinal Strain Measurements in Combination With Non-invasive ECG Parameters Predict the Success or Failure of Flecainide Treatment for Atrial Fibrillation Patients?
Brief Title: The Use of Flecainide for Treatment of Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: Tambocor_prosp_01
Record Dates: First submitted 2021-10-18; First posted 2021-10-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Global peak atrial longitudinal strain and ECG — During the follow-up period the patient will have four clinical visits, during which clinical data, advanced echocardiographic data (strain and speckle tracking) and ECGs (Glasgow criteria) will be collected

SUMMARY:
This prospective observational study will include patients with atrial fibrillation that has indication for treatement with flecainide. Included patients are followed during a 12 month period. During the follow-up period they will have four clinical visits, during which clinical data, advanced echocardiographic data (strain and speckle tracking) and ECGs (Glasgow criteria) will be collected. These data will be analysed in relation to outcome parameters as: maintaining a normal sinus rhythm (arrythmia free health status), number of AF-free months, chances of successful electrical cardioversion, frequency of side effects, risk of pro-arrhythmias and mortality. The importance of these two analyses is to improve the use of flecainide. Hence, today patients with low benefit compared to risk of adverse events are inappropriately treated with flecainide with the "trial and error" approach currently used. On the other hand flecainide is currently underutilized, and patients denied the treatment that could improve their quality of life, prognosis and reduce their risk of cardiovascular adverse events. By investigating novel and promising parameters there is the potential of a better prediction of initiating safe and accurate anti-arrhythmic therapy for patients with atrial fibrillation.

DETAILED DESCRIPTION:
Study synopsis for the Tambocor Prospective study

Inclusion: Patients with atrial fibrillation that admitted to the ward for prior to start of flecainide initiation.

Ethics: Informed Concent prior to inclusion.

Follow up after baseline: 4 visits during 12 month.

End points : Side effects that lead to discontinuation of flecainide. Persistent AF that lead to discontinuation of flecainide.

Evaluated parameters: 12 lead ECG, ECHO: LA, LV, HV strain , Dynamic Heart model: LV and RV.

The follow up visits:

Baseline: Normal ECHO after the first dose of flecainide, ECG and Questionnaire

4 Weeks: Normal ECHO + Protocol ECHO (LA, LV, HV strain , Dynamic Heart model: LV and RV) and Questionnaire.

6 month: Normal ECHO + Protocol ECHO (LA, LV, HV strain , Dynamic Heart model: LV and RV) and Questionnaire.

12 month: Normal ECHO + Protocol ECHO (LA, LV, HV strain , Dynamic Heart model: LV and RV) and Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients with written informed consent who are eligible for flecainide treatment for atrial fibrillation.
* The patients must be followed at the Skånes hospitals northwest and Skånes university hospitals.
* Age >18 years

Exclusion Criteria:

* Flecainide treatment with other indication than atrial fibrillation (including atrial flutter).
* No secure date for treatment start.
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For patients with troublesome fibrillation burden, there are about as many ways to initiate and follow up treatment with Flecainide as there are Swedish hospitals. Although it was 30 years ago that the CAST study showed that Flecainide should not be given to patients with ischemic or structural heart disease, there is a lack of knowledge about which patient characteristics predict an effective and safe treatment. Today, the clinician is forced to use Flecainide according to the "trial-and-error" method, you simply have to see which patients benefit from the drug by trying. Regardless of the effect, patients are at risk of serious proarrhythmias and side effects.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Arrythmia free health status | During the 12 month follow up
  Can we predict who will maintain a normal sinus rhythm prior to initiation of flecainide? treatment start

SECONDARY OUTCOMES:
Number of AF-free months | During the 12 month follow up
  Can we improve the number of AF-free months by a better prediction model
Frequency of side effects | During the 12 month follow up
  Can we improve the diagnostic accuracy to reduce the frequency of side effects
Risk of pro-arrhythmias | During the 12 month follow up
  Can we improve the diagnostic accuracy to reduce risk of pro-arrhythmias
Mortality | During the 12 month follow up
  Can we improve the diagnostic accuracy to reduce risk mortality

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Madsen Härdig, RN, PhD, Principal Investigator — Lund University and Region Skane
Locations (1):
- Clinical Sciences, Helsingborg Medical Faculty Lund University, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrikopoulos GK, Pastromas S, Tzeis S. Flecainide: Current status and perspectives in arrhythmia management. World J Cardiol. 2015 Feb 26;7(2):76-85. doi: 10.4330/wjc.v7.i2.76. PMID 25717355
- [Background] Aliot E, Capucci A, Crijns HJ, Goette A, Tamargo J. Twenty-five years in the making: flecainide is safe and effective for the management of atrial fibrillation. Europace. 2011 Feb;13(2):161-73. doi: 10.1093/europace/euq382. Epub 2010 Dec 7. PMID 21138930
- [Background] Cardiac Arrhythmia Suppression Trial (CAST) Investigators. Preliminary report: effect of encainide and flecainide on mortality in a randomized trial of arrhythmia suppression after myocardial infarction. N Engl J Med. 1989 Aug 10;321(6):406-12. doi: 10.1056/NEJM198908103210629. PMID 2473403
- [Background] Macfarlane PW, Devine B, Latif S, McLaughlin S, Shoat DB, Watts MP. Methodology of ECG interpretation in the Glasgow program. Methods Inf Med. 1990 Sep;29(4):354-61. PMID 2233383
- [Background] Skov MW, Ghouse J, Kuhl JT, Platonov PG, Graff C, Fuchs A, Rasmussen PV, Pietersen A, Nordestgaard BG, Torp-Pedersen C, Hansen SM, Olesen MS, Haunso S, Kober L, Gerds TA, Kofoed KF, Svendsen JH, Holst AG, Nielsen JB. Risk Prediction of Atrial Fibrillation Based on Electrocardiographic Interatrial Block. J Am Heart Assoc. 2018 May 30;7(11):e008247. doi: 10.1161/JAHA.117.008247. PMID 29848496
- [Background] Kuppahally SS, Akoum N, Burgon NS, Badger TJ, Kholmovski EG, Vijayakumar S, Rao SN, Blauer J, Fish EN, Dibella EV, Macleod RS, McGann C, Litwin SE, Marrouche NF. Left atrial strain and strain rate in patients with paroxysmal and persistent atrial fibrillation: relationship to left atrial structural remodeling detected by delayed-enhancement MRI. Circ Cardiovasc Imaging. 2010 May;3(3):231-9. doi: 10.1161/CIRCIMAGING.109.865683. Epub 2010 Feb 4. PMID 20133512